CLINICAL TRIAL: NCT00157534
Title: A Phase II, Randomised, Dose-Ranging, Open-Label, Multi-Centre Study to Evaluate the Safety and Efficacy of Celgosivir for 12 Weeks in Patients With Chronic Hepatitis C Infection
Brief Title: A Study to Evaluate the Safety and Efficacy of Celgosivir in Patients With Chronic Hepatitis C Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioWest Therapeutics Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV-04-001
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Celgosivir; HCV; Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — celgosivir

INTERVENTIONS:
Drug: Celgosivir

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of celgosivir for 12 weeks in patients with chronic hepatitis C genotype 1 infection.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 to 65 years of age, inclusive.
* Primary diagnosis of chronic HCV infection.

Exclusion Criteria:

* Patients who did not respond or relapsed following therapy with interferon.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2004-10; Study Completion 2005-08

PRIMARY OUTCOMES:
Safety analysis

SECONDARY OUTCOMES:
Hepatitis C viral load

CONTACTS AND LOCATIONS:
Overall Officials: Jim Pankovich, Study Director — BioWest Therapeutics Inc